CLINICAL TRIAL: NCT02524665
Title: U0289-404: An Evaluator Blinded, 8 Week, Split Face Study to Evaluate and Compare the Efficacy and Tolerability of MAXCLARITYII and MURAD in Subjects With Acne
Brief Title: 8 Week Study to Evaluate and Compare the Efficacy and Tolerability of MAXCLARITY II and MURAD To Treat Acne
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 114553
Record Dates: First submitted 2015-08-13; First posted 2015-08-17 (Estimated); Results first posted 2017-03-15 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-01

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Salicylic Acid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- MAXCLARITY II (Experimental): MAXCLARITY II Foam Cleanser (2.5% BPO) plus Foam Treatment (2.5% BPO) and (0.5% Salicylic Acid) Toner Foam. Available over the counter. Each subject applies both arms (MAXCLARITY II and MURAD) simultaneously for the entire duration of the study (8 weeks), each arm to be applied to one side of the face only (split-face study) according to randomization.
  Interventions: Other: MAXCLARITY II (2.5% BPO) Foam Cleanser; Other: MAXCLARITY II (2.5% BPO) Foam Treatment; Other: MAXCLARITY II (0.5% Salicylic Acid) Toner Foam
- MURAD (Active Comparator): MURADClarifying Cleanser (1.5% SA) plus Exfoliating Acne Treatment Gel (1% SA) and Skin Perfecting Lotion. Available over the counter. Each subject applies both arms (MAXCLARITY II and MURAD) simultaneously for the entire duration of the study (8 weeks), each arm to be applied to one side of the face only (split-face study) according to randomization.
  Interventions: Other: MURAD Clarifying Cleanser (1.5% SA); Other: Exfoliating Acne Treatment Gel (1% SA); Other: Skin Perfecting Lotion

INTERVENTIONS:
Other: MAXCLARITY II (2.5% BPO) Foam Cleanser — Available over the counter.
  Arms: MAXCLARITY II
Other: MAXCLARITY II (2.5% BPO) Foam Treatment — Available over the counter.
  Arms: MAXCLARITY II
Other: MAXCLARITY II (0.5% Salicylic Acid) Toner Foam — Available over the counter.
  Arms: MAXCLARITY II
Other: MURAD Clarifying Cleanser (1.5% SA) — Available over the counter.
  Arms: MURAD
Other: Exfoliating Acne Treatment Gel (1% SA) — Available over the counter.
  Arms: MURAD
Other: Skin Perfecting Lotion — Available over the counter.
  Arms: MURAD

SUMMARY:
One of the main success factors in acne therapy is user compliance with treatment, product cost, availability and ease of use. Poor compliance may translate into decreased efficacy (either not improving symptoms well enough or not improving symptoms fast enough), tolerability issues or adverse effects (eg, erythema, dryness, or peeling of the skin), a lack of understanding of the instructions for use, or product cost/availability. Whatever the reason, poor compliance translates to decreased efficacy and increased frustration on the part of the user.

The current study will evaluate and compare the efficacy and tolerability of 2 over the counter, topical product lines for the treatment of acne: MAXCLARITY II Foam Cleanser (2.5% benzoyl peroxide [BPO]) plus Foam Treatment (2.5% BPO) and (0.5% Salicylic Acid) Toner Foam compared with MURAD Clarifying Cleanser (1.5% salicylic acid [SA]) plus Exfoliating Acne Treatment Gel (1% SA) and Skin Perfecting Lotion.

DETAILED DESCRIPTION:
Acne vulgaris (acne) is an extremely common dermatological disease that is found typically in adolescence and young adulthood. Acne manifests with open and closed comedones (blackheads and whiteheads), papules, pustules, nodules, and cysts on the face, neck, and trunk. Acne can be treated with a variety of agents that are selected to address the pathogenic factors assumed to be responsible for the type and degree of manifested acne lesions. Monotherapy and combination therapy regimens are both useful. Topical agents are generally used as first-line therapy and include retinoids, antibiotic preparations (eg, erythromycin and clindamycin), benzoyl peroxide (BPO), alpha and beta hydroxy acids (eg, glycolic and salicylic acid [SA] preparations), and azelaic acid. Systemic therapies are initiated in patients with moderate to severe inflammatory acne that does not respond to topical therapy.

Benzoyl peroxide has antimicrobial and anti inflammatory properties and is often considered an important component of acne treatment. Salicylic acid has comedolytic properties and is often used when other topical therapies are not tolerated. Benzoyl peroxide and SA are frequently the first products that adolescents will use for acne because both can be purchased without a prescription in several different concentrations and formulations.

One of the main success factors in acne therapy is user compliance with treatment, product cost, availability and ease of use. Poor compliance may translate into decreased efficacy (either not improving symptoms well enough or not improving symptoms fast enough), tolerability issues or adverse effects (eg, erythema, dryness, or peeling of the skin), a lack of understanding of the instructions for use, or product cost/availability. Whatever the reason, poor compliance translates to decreased efficacy and increased frustration on the part of the user.

The current study will evaluate and compare the efficacy and tolerability of 2 over the counter, topical product lines for the treatment of acne: MAXCLARITY II Foam Cleanser (2.5% benzoyl peroxide [BPO]) plus Foam Treatment (2.5% BPO) and (0.5% Salicylic Acid) Toner Foam compared with MURADClarifying Cleanser (1.5% salicylic acid [SA]) plus Exfoliating Acne Treatment Gel (1% SA) and Skin Perfecting Lotion.

This is a randomized, single center, evaluator blinded, split face efficacy and tolerability study of MaxClarity II and Murad, 2 over the-counter, topical product lines for the treatment of acne. Approximately 20 subjects, aged from 16 to 29 years, inclusive, with mild facial acne are expected to participate in the study. No more than 50% of the subjects at each site can be enrolled under the age of 20.

An expert grader (blinded evaluator) will complete counts of inflamed lesions (papules/pustules) and noninflamed lesions (open/closed comedones), the ISGA, and an assessment of tolerability of each side of the face at each study visit. Subjects will assess tolerability on each side of the face at each study visit and will complete a product acceptability and preference questionnaire at the end of the study.

The study duration will be 8 weeks (56 days) with visits at baseline (day 1), week 1, week 2, week 4 and week 8. Only the expert grader (evaluator) will be blinded to the study product assignments; subjects and study nurses/coordinators will not be blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding and willing to provide signed and dated written voluntary informed consent (and any local or national authorization requirements) before any protocol specific procedures are performed.
2. Male or female aged from 16 to 29 years, inclusive, at time of consent. No more than 50% of the subjects at each site can be enrolled under the age of 20.
3. Mild facial acne, characterized by at least 12 facial inflammatory lesions (papules and pustules) and/or noninflammatory lesions (open and closed comedones) on each half of the face (excluding nose and front hairline areas).
4. Able to complete the study and to comply with study instructions.
5. Sexually active females of childbearing potential participating in the study must agree to use a medically acceptable method of contraception while receiving protocol-assigned product. A woman of childbearing potential is defined as one who is biologically capable of becoming pregnant; including perimenopausal women who are less than 2 years from their last menses. Acceptable contraceptive methods include the following:

   * Hormonal contraception, including oral, injectable, or implantable methods started at least 2 months prior to screening. If hormonal contraception was started less than 2 months prior to screening, then a form of nonhormonal contraception should be added until the third continuous month of hormonal contraception has been completed.
   * Two forms of reliable nonhormonal contraception, to include the use of either an intrauterine device plus a reliable barrier method or 2 reliable barrier methods. Reliable barrier methods include condoms or diaphragms. A cervical cap is also a reliable barrier method, provided that the female subject has never given birth naturally. The combined use of a condom and spermicide constitute 2 forms of acceptable nonhormonal contraception, provided that they are both used properly. The use of spermicide alone and the improper use of condoms are inferior methods of contraception. Subjects with surgical sterilization, including tubal sterilization or partner's vasectomy, must use a form of nonhormonal contraception. A barrier method or sterilization plus spermatocide is acceptable.
   * Women who are not currently sexually active must agree to use a medically accepted method of contraception should she become sexually active while participating in the study.

Exclusion Criteria:

1. Female who is pregnant, trying to become pregnant, or breast feeding.
2. Has an active or chronic skin allergy.
3. Has a history of acute or chronic disease that might interfere with or increase the risk of study participation.
4. Had skin cancer treatment in preceding 12 months.
5. Has damaged skin on facial areas (eg, sunburn, tattoo, or scar)
6. Had any medical procedure (eg, laser resurfacing, chemical peel, or plastic surgery) on facial areas in preceding 12 months.
7. Had any cosmetic procedure (eg, microdermabrasion) on facial areas within 8 weeks of the baseline visit.
8. Has any dermatological disorder that in the opinion of the investigator may interfere with the accurate evaluation of the subject's facial appearance.
9. Received any investigational drug or procedure within 28 days of the baseline visit.
10. Currently using any medication that in the opinion of the investigator may affect the evaluation of the study products or place the subject at undue risk.
11. Has a history of known or suspected intolerance to any of the ingredients of the study products (ie, benzoyl peroxide).
12. Considered unable or unlikely to attend the necessary visits.
13. Live in the same household as currently enrolled subjects.
14. Employee of the investigator, a contract research organization, or Stiefel Laboratories who is involved in the study, or an immediate family member (partner, offspring, parents, siblings or sibling's offspring) of an employee involved in the study.

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2009-09; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 114553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 114553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 114553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 114553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 114553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 114553 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From September-2009 to December-2009, total 20 participants were randomized at one of center in Louisville. MAXCLARITY II™ is a trademark of Stiefel Laboratories, Inc and MURAD™ is licensed product of Murad Europe Limited.
Pre-assignment Details: Male or female participants 18 to 29 years of age with mild facial acne vulgaris, characterized by at least 24 facial inflammatory lesions (papules and pustules) and/or non-inflammatory lesions (open and closed comedones) on each half of the face (excluding nose and front hairline areas) were included.
Groups:
- MAXCLARITY II + Murad: MaxClarity II was a 2.5 percent (%) benzoyl peroxide (BPO) foam cleanser and foam treatment, 0.5% salicylic acid (SA) toner foam. Murad clarifying cleanser was a 1.5% SA plus exfoliating acne treatment gel (1% SA) and skin perfecting lotion. Both treatments were applied topically to 1 side of face twice daily (BD) for 8 weeks. MaxClarity II application: Participants washed the assigned side of face with the foam cleanser, patted dry twice and then applied foam treatment in ante meridiem (AM) and toner foam in post meridiem (PM). Murad application: In first week of treatment, participants washed the assigned side of face with the clarifying cleanser, patted dry twice and applied acne treatment gel, then applied skin perfecting lotion in AM and skin perfecting lotion only in PM. During weeks 2-8, in AM and PM, participants washed assigned side of the face with clarifying cleanser, patted dry, applied acne treatment gel, then applied skin perfecting lotion.
Period: Overall Study
Arm/Group | MAXCLARITY II + Murad
Started | 20
Completed | 19
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | MAXCLARITY II + Murad
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.5 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 10
Race/Ethnicity, Customized [Number; unit: Participants]
  Black | 7
  White | 13

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change in Inflammatory, Non-inflammatory and Total Lesion Counts From Baseline to Week 8.
Description: During each study visit, expert grader (blinded evaluator) assessed the left side and right side of the face as inflammatory (papules [solid elevation of skin with no visible fluid] and pustules [small inflamed elevation of the skin that is filled with pus]) and non-inflammatory (open [blackheads] and closed [whiteheads] comedones) and total lesions for each participant. Each type of lesion was counted separately; the lesion counts were taken from the face from hairline to the mandible (including forehead, cheeks, and chin). Total lesion counts were calculated as the sum of the inflammatory and non-inflammatory lesion counts. Percent change from Baseline to Week 8 was calculated as the value at Week 8 minus the value at Baseline divided by the Baseline value multiplied by 100. Baseline is defined as value at Day 1.
Time Frame: Baseline and Week 8
Population: Intent-to-treat (ITT) analysis set was used which included data from all randomized participants who received study product. Only those participants available at the specified time points were analyzed (represented by n=X,X in the category titles).
Measure: Mean (Standard Deviation); unit: Percent change
Groups:
- MAXCLARITY II: MAXCLARITY II was a 2.5% BPO foam cleanser and foam treatment, 0.5% SA toner foam. It was applied topically to 1 side of face BD for 8 weeks. Participants washed the assigned side of face with the foam cleanser, patted dry twice and then applied foam treatment in AM and toner foam in PM.
- Murad: Murad clarifying cleanser was a 1.5% SA plus exfoliating acne treatment gel (1% SA) and skin perfecting lotion. It was applied topically to 1 side of face BD for 8 weeks. In first week of treatment, participants washed the assigned side of face with the clarifying cleanser, patted dry twice and applied acne treatment gel, then applied skin perfecting lotion in AM and skin perfecting lotion only in PM. During weeks 2-8, in AM and PM, participants washed assigned side of the face with clarifying cleanser, patted dry, applied acne treatment gel, then applied skin perfecting lotion.
Arm/Group | MAXCLARITY II | Murad
Number analyzed (Participants) | 20 | 20
Percent change
  Inflammatory lesion counts- Week 8, n=19, 17 | -78.70 (40.93) | -61.52 (47.59)
  Non-inflammatory lesion counts- Week 8, n=19, 19 | -69.32 (48.69) | -77.09 (23.50)
  Total lesion counts-Week 8, n=19, 19 | -76.67 (30.79) | -75.01 (23.22)
Statistical Analysis 1: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.0769, Wilcoxon signed-rank test — The assumption of normality was verified using a Shapiro-Wilk Test. If the assumption of normality was rejected (at the 0.01 level), a non-parametric method (Wilcoxon signed-rank test) was used; Mean Difference (Final Values) = -14.67, Standard Deviation 61.97 — Comparison of inflammatory lesion counts between MAXCLARITY II and Murad at Week 8
Statistical Analysis 2: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.6698, Wilcoxon signed-rank test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.77, Standard Deviation 33.73 — Comparison of non-inflammatory lesion counts between MAXCLARITY II and Murad at Week 8
Statistical Analysis 3: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.6854, t-test, 2 sided — Percent change from baseline were analyzed using the individual differences between both sides of the face at an alpha level of 0.05 using paired t-tests; Mean Difference (Final Values) = -1.66, Standard Deviation 17.59 — Comparison of total lesion counts between MAXCLARITY II and Murad at Week 8

2. Secondary Outcome: Mean Percent Change in Inflammatory, Non-inflammatory and Total Lesion Counts From Baseline to Week 1, 2 and 4.
Description: During each study visit, expert grader (blinded evaluator) assessed the left side and right side of the face as inflammatory (papules [solid elevation of skin with no visible fluid] and pustules [small inflamed elevation of the skin that is filled with pus]) and non-inflammatory (open comedones [blackheads] and closed comedones [whiteheads]) and total lesions for each participant. Each type of lesion was counted separately; the lesion counts were taken from the face from hairline to the mandible (including forehead, cheeks, and chin). Total lesion counts were calculated as the sum of the inflammatory and non-inflammatory lesion counts. Percent change from Baseline to scheduled time point was calculated as the value at scheduled time point minus the value at Baseline divided by the Baseline value multiplied by 100. Baseline is defined as value at Day 1.
Time Frame: Baseline and Week 1, 2, 4
Population: ITT analysis set. Only those participants available at the specified time points were analyzed (represented by n=X,X in the category titles).
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | MAXCLARITY II | Murad
Number analyzed (Participants) | 20 | 20
Percent change
  Inflammatory lesion counts- Week 1, n=19, 17 | -17.69 (38.89) | -7.85 (83.21)
  Inflammatory lesion counts- Week 2, n=19, 17 | -46.69 (55.00) | -14.25 (66.06)
  Inflammatory lesion counts- Week 4, n=19, 17 | -55.35 (46.13) | -51.95 (47.60)
  Non-inflammatory lesion counts- Week 1, n=19, 19 | -4.94 (52.60) | -15.92 (28.91)
  Non-inflammatory lesion counts- Week 2, n=19, 19 | -28.07 (48.27) | -37.07 (28.42)
  Non-inflammatory lesion counts- Week 4, n=19, 19 | -52.85 (47.46) | -60.27 (24.54)
  Total lesion counts-Week 1, n=19, 19 | -12.57 (27.27) | -18.29 (23.53)
  Total lesion counts-Week 2, n=19, 19 | -37.06 (27.97) | -35.84 (22.91)
  Total lesion counts-Week 4, n=19, 19 | -60.93 (26.94) | -60.73 (22.49)
Statistical Analysis 1: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.5031, Wilcoxon signed-rank test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.10, Standard Deviation 74.55 — Comparison of percent change inflammatory lesion counts between MAXCLARITY II and Murad at Week 1
Statistical Analysis 2: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.2464, t-test, 2 sided — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = -29.11, Standard Deviation 99.76 — Comparison of percent change inflammatory lesion counts between MAXCLARITY II and Murad at Week 2
Statistical Analysis 3: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.8894, Wilcoxon signed-rank test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -4.03, Standard Deviation 65.22 — Comparison of percent change inflammatory lesion counts between MAXCLARITY II and Murad at Week 4
Statistical Analysis 4: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.6722, Wilcoxon signed-rank test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 10.98, Standard Error of Mean 46.04 — Comparison of percent change non-inflammatory lesion counts between MAXCLARITY II and Murad at Week 1
Statistical Analysis 5: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.3352, t-test, 2 sided — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 8.99, Standard Deviation 39.59 — Comparison of percent change non-inflammatory lesion counts between MAXCLARITY II and Murad at Week 2
Statistical Analysis 6: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.9323, Wilcoxon signed-rank test — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.41, Standard Deviation 35.46 — Comparison of percent change non-inflammatory lesion counts between MAXCLARITY II and Murad at Week 4
Statistical Analysis 7: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.3513, t-test, 2 sided — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = 5.72, Standard Deviation 26.05 — Comparison of percent change total lesion counts between MAXCLARITY II and Murad at Week 1
Statistical Analysis 8: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.8199, t-test, 2 sided — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = -1.22, Standard Deviation 22.97 — Comparison of percent change total lesion counts between MAXCLARITY II and Murad at Week 2
Statistical Analysis 9: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.9616, t-test, 2 sided — [p-value comment as in outcome 1, analysis 3]; Mean Difference (Final Values) = -0.20, Standard Deviation 17.83 — Comparison of percent change total lesion counts between MAXCLARITY II and Murad at Week 4

3. Secondary Outcome: Mean Change in Investigator's Static Global Assessment (ISGA) From Baseline to Week 1, 2, 4 and 8
Description: During each study visit, investigators/expert grader evaluated the acne severity of participants' faces using the ISGA scale on right and left side of face on a five point scale from 0 to 4 defined as 0-clear, 1-almost clear, 2-mild, 3-moderate, 4-severe. Change from Baseline to scheduled time point was calculated as the value at scheduled time point minus the value at Baseline. Baseline is defined as value at Day 1.
Time Frame: Baseline and Week 1, 2, 4, 8
Population: ITT analysis set. Only those participants available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MAXCLARITY II | Murad
Number analyzed (Participants) | 19 | 19
Score on a scale
  ISGA score-Week 1 | -0.05 (0.40) | -0.11 (0.32)
  ISGA score -Week 2 | -0.16 (0.60) | -0.05 (0.40)
  ISGA score -Week 4 | -0.47 (0.70) | -0.58 (0.51)
  ISGA score -Week 8 | -1.16 (0.90) | -0.89 (0.74)
Statistical Analysis 1: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test; Mean Difference (Final Values) = 0.05, Standard Deviation 0.23 — Comparison of ISGA score between MAXCLARITY II and Murad at Week 1
Statistical Analysis 2: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.7500, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.11, Standard Deviation 0.66 — Comparison of ISGA score between MAXCLARITY II and Murad at Week 2
Statistical Analysis 3: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.7539, Wilcoxon signed-rank test; Mean Difference (Final Values) = 0.11, Standard Deviation 0.74 — Comparison of ISGA score between MAXCLARITY II and Murad at Week 4
Statistical Analysis 4: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.3071, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.26, Standard Deviation 0.87 — Comparison of ISGA score between MAXCLARITY II and Murad at Week 8

4. Secondary Outcome: Change in Investigator Assessment of Tolerability (Erythema, Dryness and Peeling) From Baseline to Weeks 1, 2, 4 and 8.
Description: Erythema (redness), dryness, and peeling, were evaluated independently by the investigator on a five point scale from 0 to 4 defined as 0-none, 1-very minimal, 2-mild, 3-moderate, 4-severe. Change from Baseline to scheduled time point was calculated as the value at scheduled time point minus the value at Baseline. Baseline is defined as value at Day 1.
Time Frame: Baseline and Week 1, 2, 4, 8
Population: ITT analysis set. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MAXCLARITY II | Murad
Number analyzed (Participants) | 19 | 19
Score on a scale
  Erythema score-Week 1 | 0.16 (0.83) | 0.00 (0.67)
  Erythema score -Week 2 | -0.21 (0.54) | -0.16 (0.76)
  Erythema score -Week 4 | -0.37 (0.83) | -0.32 (0.89)
  Erythema score -Week 8 | -0.32 (1.06) | -0.32 (1.06)
  Dryness score-Week 1 | 0.11 (0.81) | 0.00 (0.33)
  Dryness score -Week 2 | -0.11 (0.32) | -0.11 (0.32)
  Dryness score -Week 4 | -0.05 (0.40) | -0.05 (0.40)
  Dryness score -Week 8 | 0.00 (0.47) | 0.05 (0.52)
  Peeling score-Week 1 | 0.05 (0.78) | -0.11 (0.32)
  Peeling score -Week 2 | -0.11 (0.32) | -0.11 (0.32)
  Peeling score -Week 4 | -0.05 (0.40) | -0.05 (0.40)
  Peeling score -Week 8 | -0.11 (0.32) | -0.05 (0.40)
Statistical Analysis 1: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.5000, Wilcoxon signed-rank test; Mean Difference (Final Values) = 0.16, Standard Deviation 0.50 — Comparison of Erythema score between MAXCLARITY II and Murad at Week 1
Statistical Analysis 2: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.05, Standard Deviation 0.52 — Comparison of Erythema score between MAXCLARITY II and Murad at Week 2
Statistical Analysis 3: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.05, Standard Deviation 0.23 — Comparison of Erythema score between MAXCLARITY II and Murad at Week 4
Statistical Analysis 4: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0, Wilcoxon signed-rank test — The value is mentioned as '0', as no P-value generated; Mean Difference (Final Values) = 0.00, Standard Deviation 0.00 — Comparison of Erythema score between MAXCLARITY II and Murad at Week 8
Statistical Analysis 5: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test; Mean Difference (Final Values) = 0.11, Standard Deviation 0.74 — Comparison of Dryness score between MAXCLARITY II and Murad at Week 1
Statistical Analysis 6: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0, Wilcoxon signed-rank test — The value is mentioned as '0', as no P-value generated; Mean Difference (Final Values) = 0.00, Standard Deviation 0.00 — Comparison of Dryness score between MAXCLARITY II and Murad at Week 2
Statistical Analysis 7: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0, Wilcoxon signed-rank test — The value is mentioned as '0', as no P-value generated; Mean Difference (Final Values) = 0.00, Standard Deviation 0.00 — Comparison of Dryness score between MAXCLARITY II and Murad at Week 4
Statistical Analysis 8: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.05, Standard Deviation 0.23 — Comparison of Dryness score between MAXCLARITY II and Murad at Week 8
Statistical Analysis 9: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test; Mean Difference (Final Values) = 0.16, Standard Deviation 0.69 — Comparison of Peeling score between MAXCLARITY II and Murad at Week 1
Statistical Analysis 10: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0, Wilcoxon signed-rank test — The value is mentioned as '0', as no P-value generated; Mean Difference (Final Values) = 0.00, Standard Deviation 0.00 — Comparison of Peeling score between MAXCLARITY II and Murad at Week 2
Statistical Analysis 11: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0, Wilcoxon signed-rank test — The value is mentioned as '0', as no P-value generated; Mean Difference (Final Values) = 0.00, Standard Deviation 0.00 — Comparison of Peeling score between MAXCLARITY II and Murad at Week 4
Statistical Analysis 12: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.05, Standard Deviation 0.23 — Comparison of Peeling score between MAXCLARITY II and Murad at Week 8

5. Secondary Outcome: Change in Participant Assessment of Tolerability (Redness, Dryness, Burning, Itching and Scaling) From Baseline to Weeks 1, 2, 4 and 8.
Description: Redness, dryness, burning, itching and scaling were evaluated independently by the participant on a five point scale from 0 to 4 defined as 0-none, 1-very minimal, 2-mild, 3-moderate, 4-severe. Change from Baseline to scheduled time point was calculated as the value at scheduled time point minus the value at Baseline. Baseline is defined as value at Day 1.
Time Frame: Baseline and Week 1, 2, 4, 8
Population: ITT analysis set. Only those participants with data available at the indicated time points were analyzed.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | MAXCLARITY II | Murad
Number analyzed (Participants) | 19 | 19
Score on a scale
  Redness score-Week 1 | -0.11 (0.88) | -0.32 (0.48)
  Redness score -Week 2 | -0.11 (0.81) | -0.26 (0.56)
  Redness score -Week 4 | -0.32 (0.58) | -0.11 (1.15)
  Redness score -Week 8 | -0.42 (0.69) | -0.26 (1.05)
  Dryness score-Week 1 | -0.21 (1.47) | -0.11 (1.20)
  Dryness score -Week 2 | -0.16 (1.46) | -0.26 (0.93)
  Dryness score -Week 4 | -0.37 (1.21) | -0.11 (1.49)
  Dryness score -Week 8 | -0.42 (1.22) | -0.11 (1.52)
  Burning score-Week 1 | 0.11 (1.15) | 0.16 (1.12)
  Burning score -Week 2 | -0.11 (0.57) | 0.00 (0.88)
  Burning score -Week 4 | -0.26 (0.65) | -0.05 (0.91)
  Burning score -Week 8 | -0.26 (0.87) | 0.00 (0.82)
  Itching score-Week 1 | -0.21 (0.71) | 0.00 (0.88)
  Itching score -Week 2 | 0.00 (0.88) | 0.11 (0.94)
  Itching score -Week 4 | -0.26 (0.87) | 0.11 (1.24)
  Itching score -Week 8 | -0.21 (0.63) | 0.11 (1.10)
  Scaling score-Week 1 | 0.05 (1.18) | -0.11 (1.05)
  Scaling score -Week 2 | -0.26 (0.87) | -0.26 (0.87)
  Scaling score -Week 4 | -0.16 (1.12) | 0.11 (1.49)
  Scaling score -Week 8 | 0.11 (0.94) | 0.21 (1.08)
Statistical Analysis 1: Comparison: MAXCLARITY II; Test type: Superiority or Other; p = 0.5000, Wilcoxon signed-rank test; Mean Difference (Final Values) = 0.21, Standard Deviation 0.63 — Comparison of Redness score between MAXCLARITY II and Murad at Week 1
Statistical Analysis 2: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.5000, Wilcoxon signed-rank test; Mean Difference (Final Values) = 0.16, Standard Deviation 0.50 — Comparison of Redness score between MAXCLARITY II and Murad at Week 2
Statistical Analysis 3: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.21, Standard Deviation 0.92 — Comparison of Redness score between MAXCLARITY II and Murad at Week 4
Statistical Analysis 4: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.16, Standard Deviation 0.69 — Comparison of Redness score between MAXCLARITY II and Murad at Week 8
Statistical Analysis 5: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.8125, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.11, Standard Deviation 0.88 — Comparison of Dryness score between MAXCLARITY II and Murad at Week 1
Statistical Analysis 6: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.5742, Wilcoxon signed-rank test; Mean Difference (Final Values) = 0.11, Standard Deviation 0.94 — Comparison of Dryness score between MAXCLARITY II and Murad at Week 2
Statistical Analysis 7: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.5000, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.26, Standard Deviation 0.93 — Comparison of Dryness score between MAXCLARITY II and Murad at Week 4
Statistical Analysis 8: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.2500, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.32, Standard Deviation 0.82 — Comparison of Dryness score between MAXCLARITY II and Murad at Week 8
Statistical Analysis 9: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.05, Standard Deviation 0.62 — Comparison of Burning score between MAXCLARITY II and Murad at Week 1
Statistical Analysis 10: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.7500, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.11, Standard Deviation 0.74 — Comparison of Burning score between MAXCLARITY II and Murad at Week 2
Statistical Analysis 11: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.7500, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.21, Standard Deviation 0.98 — Comparison of Burning score between MAXCLARITY II and Murad at Week 4
Statistical Analysis 12: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.2500, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.26, Standard Deviation 0.73 — Comparison of Burning score between MAXCLARITY II and Murad at Week 8
Statistical Analysis 13: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.2500, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.21, Standard Deviation 0.54 — Comparison of Itching score between MAXCLARITY II and Murad at Week 1
Statistical Analysis 14: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.7500, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.11, Standard Deviation 0.74 — Comparison of Itching score between MAXCLARITY II and Murad at Week 2
Statistical Analysis 15: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.2500, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.37, Standard Deviation 1.01 — Comparison of Itching score between MAXCLARITY II and Murad at Week 4
Statistical Analysis 16: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.2500, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.32, Standard Deviation 0.82 — Comparison of Itching score between MAXCLARITY II and Murad at Week 8
Statistical Analysis 17: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.5000, Wilcoxon signed-rank test; Mean Difference (Final Values) = 0.16, Standard Deviation 0.50 — Comparison of Scaling score between MAXCLARITY II and Murad at Week 1
Statistical Analysis 18: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0, Wilcoxon signed-rank test — The value is mentioned as '0', as no P-value generated; Mean Difference (Final Values) = 0.00, Standard Deviation 0.00 — Comparison of Scaling score between MAXCLARITY II and Murad at Week 2
Statistical Analysis 19: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.5000, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.26, Standard Deviation 0.93 — Comparison of Scaling score between MAXCLARITY II and Murad at Week 4
Statistical Analysis 20: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, Wilcoxon signed-rank test; Mean Difference (Final Values) = -0.11, Standard Deviation 0.81 — Comparison of Scaling score between MAXCLARITY II and Murad at Week 8

6. Secondary Outcome: Percentage of Participant Who Improved by at Least One Grade on the ISGA
Description: During each study visit, investigators/expert grader evaluated the acne severity of participants' faces using the ISGA scale on right and left side of face on a five point scale from 0 to 4 defined as 0-clear, 1-almost clear, 2-mild, 3-moderate, 4-severe. Percent change from Baseline to scheduled time point was calculated as the value at scheduled time point minus the value at Baseline divided by the Baseline value multiplied by 100. Baseline is defined as value at Day 1.
Time Frame: Up to Week 8
Population: ITT analysis set. Only those participants with data available at the indicated time points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | MAXCLARITY II | Murad
Number analyzed (Participants) | 19 | 19
Percentage of participants
  One or more grade improvement-Week 1 | 10.5 | 10.5
  Two or more grade improvement-Week 1 | 0.0 | 0.0
  One or more grade improvement-Week 2 | 15.8 | 10.5
  Two or more grade improvement-Week 2 | 5.3 | 0.0
  One or more grade improvement-Week 4 | 47.4 | 57.9
  Two or more grade improvement-Week 4 | 5.3 | 0.0
  One or more grade improvement-Week 8 | 78.9 | 68.4
  Two or more grade improvement-Week 8 | 42.1 | 21.1
Statistical Analysis 1: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, McNemar — Comparison of one or more grade improvement between MAXCLARITY II and Murad at Week 1
Statistical Analysis 2: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0, McNemar — The value is mentioned as '0', as no P-value generated. Comparison of two or more grade improvement between MAXCLARITY II and Murad at Week 1
Statistical Analysis 3: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.5637, McNemar — Comparison of one or more grade improvement between MAXCLARITY II and Murad at Week 2
Statistical Analysis 4: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, McNemar — Comparison of two or more grade improvement between MAXCLARITY II and Murad at Week 2
Statistical Analysis 5: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.4795, McNemar — Comparison of one or more grade improvement between MAXCLARITY II and Murad at Week 4
Statistical Analysis 6: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 1.0000, McNemar — Comparison of two or more grade improvement between MAXCLARITY II and Murad at Week 4
Statistical Analysis 7: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.3173, McNemar — Comparison of one or more grade improvement between MAXCLARITY II and Murad at Week 8
Statistical Analysis 8: Comparison: MAXCLARITY II vs Murad; Test type: Superiority or Other; p = 0.1573, McNemar — Comparison of two or more grade improvement between MAXCLARITY II and Murad at Week 8

ADVERSE EVENTS:
Time Frame: Adverse events (AE) and serious adverse events (SAE) were reported through out the study (up to Week 8)
Description: An AE was an unintended or unfavorable sign, symptoms or disease, can include lack of efficacy, abuse or misuse. The SAE was an AE that results in death, life threatening, persistent or significant disability/incapacity, results in or prolongs inpatient hospitalization, congenital abnormality or birth defect. ITT analysis set used.
Arm/Group | MAXCLARITY II + Murad
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 10/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MAXCLARITY II + Murad (N=20)
Nasopharyngitis (Infections and infestations) | 3
Influenza (Infections and infestations) | 2
Body tinea (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1
Tooth caries (Gastrointestinal disorders) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Paraesthesia (Nervous system disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Endodontic procedure (Surgical and medical procedures) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.